CLINICAL TRIAL: NCT00439621
Title: A Randomized, Double-Blind, Placebo-Controlled Safety and Tolerability Study of Repeated Doses of Anti-IgE Immunotherapy in Allergic Patients
Brief Title: Safety Study of Anti-IgE Immunotherapy in Allergic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Resistentia Pharmaceuticals AB (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-24
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Allergy
Keywords: immunotherapy; allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Biological: RP 01
- 2 (Experimental)
  Interventions: Biological: RP 01
- 3 (Experimental)
  Interventions: Biological: RP 01
- 4 (Placebo Comparator)
  Interventions: Biological: RP 01

INTERVENTIONS:
Biological: RP 01 — Active immunotherapy

SUMMARY:
The purpose of the study is to evaluate safety and efficacy of three doses and two dosing regimens of RP01 as an anti-IgE immunotherapy in allergic patients.

DETAILED DESCRIPTION:
Immunotherapy is based on the principle of eliciting an immune reaction in order to block the negative effect of a specific disease-causing protein. The potential to treat diseases by means of immunotherapy instead of using conventional drugs represents an attractive opportunity in a number of chronic disease areas, including asthma and allergy. Resistentia's model to treat allergic diseases, and ultimately asthma, is to use the immune system to produce antibodies against the IgE molecules themselves. The resulting anti-IgE antibodies intercept and form complexes with the IgE molecules before they can bind to the mast cells and basophils and are thus able to block any allergen-triggered inflammatory reaction. The approach works in all types of IgE-mediated allergies independently of allergen, and also in patients sensitive to multiple allergens.

Comparisons: Three doses and two dosing regimes of RP01 will be compared as regards safety and effect.

ELIGIBILITY:
Inclusion Criteria:

* Allergy to at least one aero allergen
* Increased serum IgE level

Exclusion Criteria:

* Diagnosis of asthma
* Recent use of systemic corticosteroids or immunosuppressive treatment
* Allergy vaccination therapy

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 0-12 months

SECONDARY OUTCOMES:
Immune kinetic parameters | 0-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vidar Wendel-Hansen, MD, PhD, Study Director — Resistentia Pharmaceuticals AB
Locations (2):
- New Zealand (2):
  - P3 Research, Tauranga
  - P3 Research, Wellington